CLINICAL TRIAL: NCT03560609
Title: Optic Nerve Head Structural Response to IOP Elevation in Patients With Keratoconus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated due to the departure of the Principal Investigator from the Sponsoring institution.
Sponsor: NYU Langone Health (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01360; R01EY013178 (NIH)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Keratoconus; Glaucoma
MeSH Terms: conditions — Keratoconus; Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Subjects With Keratoconus (Active Comparator)
  Interventions: Device: Ophthalmodynamometer; Device: Goldmann applanation tonometer; Device: Pentacam; Device: ORA; Device: Optical Coherence Tomography (OCT)
- Subjects with Glaucoma (Active Comparator)
  Interventions: Device: Ophthalmodynamometer; Device: Goldmann applanation tonometer; Device: Pentacam; Device: ORA; Device: Optical Coherence Tomography (OCT)

INTERVENTIONS:
Device: Ophthalmodynamometer — The ODM (Baillart ophthlmodynamometer) is a disc attached to a piston that induces a controlled force on a fixed area. The device will be used to apply a pressure within the range of 10 mmHg - 50 mmHg 4 times to each eye. Each increase of pressure will last approximately 30 seconds. The device is FDA approved and will be used as routinely used in clinical practice
Device: Goldmann applanation tonometer — The Goldmann applanation tonometer (Haag-Streit, Basel, Switzerland) measures the IOP after the eye is numbed with a drop of anesthetic (proparacaine), which is approved by the FDA. Proparacaine is part of routine patient care using a tonometer regardless of participation in this study. The instrument's tip lightly touches the surface of the cornea and the IOP is measured. The device is FDA approved is routinely used in clinical practice.
Device: Pentacam — This device maps the cornea and provides pachymetry, topography and corneal aberration maps. The device is FDA approved and routinely used in clinical practice.
Device: ORA — ORA is an air puff tonometer that applies controlled force to flattens the cornea and provides the corneal hysteresis and corneal resistance factor. The device is FDA approved and routinely used in clinical practice.
Device: Optical Coherence Tomography (OCT) — OCT is a non-contact,real-time, high resolution, and reproducible imaging modality that provides in-vivo optical cross-sectional scanning of the retina, the ONH and of the anterior segment structures including the cornea. Clinical staff will perform subject testing, not research coordinators. Information about these non-FDA approved OCTs and the multi-modal adaptive optics system can be found in appendices A, B, C, and D. With all devices, the participant sits in a slit lamp like frame. A low power laser light is projected toward the back of their eyes while the subject fixates on a target. None of the systems produce harmful radioactive radiation.

SUMMARY:
The mechanism by which vision loss in glaucoma occurs is still unknown, but it is clear that increased Intraocular Pressure (IOP) is a major risk factor. It is also thought that the lamina cribrosa (LC) is a site of primary damage during the pathogenesis of the disease. The changes caused by intraocular pressure (IOP) modulation at the level of the optic nerve head and LC will be evaluated in the present study. Subjects with keratoconus exhibit abnormal collagen properties that can impair their LC behavior. By evaluating their lamina biomechanical response we can advance our understanding on the role of the lamina in glaucoma pathogenesis. A better understanding of the process will ultimately lead to improved detection and management of glaucoma.

It is hypothesized that subjects with keratoconus have an abnormal biomechanical response of the lamina cribrosa in response to IOP modulation.

ELIGIBILITY:
Inclusion Criteria:

Candidates must meet the following inclusion criteria in order to participate in the study.

* Ability to provide informed consent and to understand the study procedures

Keratoconus:

* Clinical diagnosis of keratoconus
* Central thinning of the cornea
* Abnormal posterior ectasia.

Glaucoma:

* Glaucomatous ONH abnormality: rim thinning, notching, undermining (excavation) or diffuse or localized RNFL defects that are characteristic of glaucoma.
* Two consecutive abnormal SITA standard perimetry tests with GHT outside normal limits.

Exclusion Criteria:

Candidates that meet any of the exclusion criteria at baseline will be excluded from study participation.

* Media opacity (e.g. lens, vitreous, cornea).
* Strabismus, nystagmus or a condition that would prevent fixation.
* Diabetes with evidence of retinopathy.
* Previous intraocular surgery or ocular trauma (with the exception of laser procedures and subjects that have undergone uneventful cataract surgery more than 6 months from enrollment date).
* Neurological and non-glaucomatous causes for visual field damage.
* Any intraocular non-glaucomatous ocular disorders.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Wollstein, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Data is available upon reasonable request indefinitely
Access Criteria: Requests should be directed to Gadi.wollstein@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated due to the departure of the Principal Investigator from the Sponsoring institution. 3 participants were enrolled in the study; none of these participants were assessed for outcome measures. No participants (n=0) were enrolled into the "Subjects with Glaucoma" arm.
Groups:
- Subjects With Keratoconus: Individuals with keratoconus.
- Subjects With Glaucoma: Individuals with glaucoma.
Period: Overall Study
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Study terminated due to departure of Principal Investigator from Sponsoring institution | 3 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated due to the departure of the Principal Investigator from the Sponsoring institution. No participants (n=0) were enrolled into the "Subjects with Glaucoma" arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.66 (4.714) |  | 38.66 (4.714)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 2 |  | 2
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Tissue Deformation in ONH Region
Description: Determination of tissue deformation will be obtained from OCT images.
Time Frame: 1 Day
Population: This study was terminated due to the departure of the Principal Investigator from the Sponsoring institution. N=3 participants were enrolled in the study in the "Subjects with Keratoconus" arm, N=0 participants were enrolled in the "Subjects with Glaucoma". N=0 participants were assessed for outcome measures prior to study closure.
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Patients With Tissue Deformation in Peripapillary Region
Description: Determination of tissue deformation will be obtained from OCT images.
Time Frame: 1 Day
Population: as for outcome 1
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Rim Area (ONH Region) Under Elevated Intraocular Pressure
Description: Obtained via OCT images - measure is from baseline to time of measurement during administration of elevated intraocular pressure.
Time Frame: 1 Day
Population: as for outcome 1
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Rim Area (Peripapillary Region) Under Elevated Intraocular Pressure
Description: as for outcome 3
Time Frame: 1 Day
Population: as for outcome 1
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change in Cup Depth (ONH Region) Under Elevated Intraocular Pressure
Description: as for outcome 3
Time Frame: 1 Day
Population: as for outcome 1
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change in Cup Depth (Peripapillary Region) Under Elevated Intraocular Pressure
Description: as for outcome 3
Time Frame: 1 Day
Population: as for outcome 1
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Change in Lamina Cibrosa Area (ONH Region) Under Elevated Intraocular Pressure
Description: as for outcome 3
Time Frame: 1 Day
Population: as for outcome 1
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Change in Lamina Cibrosa Area (Peripapillary Region) Under Elevated Intraocular Pressure
Description: as for outcome 3
Time Frame: 1 Day
Population: as for outcome 1
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day of collection of baseline characteristic data - 1 day)
Description: No participants (n=0) were enrolled into the "Subjects with Glaucoma" arm.
Arm/Group | Subjects With Keratoconus | Subjects With Glaucoma
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT03560609/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03560609/ICF_001.pdf